CLINICAL TRIAL: NCT02990039
Title: A Tailored Feasibility Study to Increase Physical Activity and to Reduce Sedentary Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FKZ 81Z5400152
Record Dates: First submitted 2016-11-15; First posted 2016-12-12 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Risk Factor
Keywords: physical activity; sedentary time; feasibility study; accelerometer
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling letter (intervention group) (Experimental): Participants of the intervention group received a brief counseling letter intervention aiming to reduce sedentary time and to increase physical activity. The intervention comprised up to three tailored letters based on separate questionnaires.
  Interventions: Behavioral: Counseling letter
- No counseling letter (control group) (No Intervention): Participants of the control group did not received the brief counseling letter intervention.

INTERVENTIONS:
Behavioral: Counseling letter — The intervention is based on the Health Action Process Approach. The first letter provides information on knowledge regarding sedentary time and physical activity as well as intervenes on self-efficacy depending on the mindset of participants (non-intender, intender, actor). The second letter focuses on benefits and barriers of physical activity as well as the role of social support for physical activity. In case of actional stage, the third letter intervenes on self-efficacy again and suggests action and coping planning. Otherwise, the letter includes ipsative feedback according to the second letter.
  Other Names: Feasibility of brief counseling letter intervention
  Arms: Counseling letter (intervention group)

SUMMARY:
The purpose of this study was (i) to develop a brief counseling letter intervention aiming to reduce sedentary time and to increase physical activity during leisure time among adults aged 42 to 64 years and (ii) to provide information on the feasibility.

DETAILED DESCRIPTION:
The study aimed to assess the feasibility of a brief counseling letter intervention to increase physical activity and to reduce sedentary time in leisure time.

Following the Intervention Mapping Protocol we developed the counseling letter intervention. The intervention is based on the Health Action Process Approach, comprising 3 tailored letters based on separate assessments, delivered over 6 month.

All participants consented (i) to participate in an examination at the university hospital including standardized measurements of blood pressure, waist and hip circumference, body height and weight as well as blood sample taking, (ii) to fill in a paper-pencil questionnaire, and (iii) to wear an accelerometer for 7 days at baseline and at 12-month follow-up.

A general population sample of cardiovascular healthy adults was randomly allocated to a control and an intervention group. At 5 time points (baseline, 3-month, 6-month, 7-month, and 12-month follow-up) participants of both study groups completed standardized questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* age between 42 and 65 years
* resident in a pre-defined zip-code area

Exclusion Criteria:

* cardiovascular event (myocardial infarction, stroke) or vascular intervention
* self-reported body-mass-index over 35 kg/m²

Ages: 42 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Adherence: Drop-out rates in control and intervention group | up to 12 month
  Measures: Analyses of drop-out rates (%) in control and intervention group

SECONDARY OUTCOMES:
Feasibility: Comprehensibility on intervention material via paper-pencil-assessment | 12 month
  Measures: questions regarding the comprehensibility on intervention material (via paper-pencil-assessment)
physical activity by self-report | Change from Baseline Physical Activity at 12 months
  Measures: paper-pencil-assessment (International Physical Activity Questionnaire-Long version, IPAQ-L)
physical activity by accelerometry | Change from Baseline Physical Activity at 12 months
  Measures: objective measurement of physical activity by accelerometry
sedentary time by self-report | Change from Baseline Sedentary Time at 12 months
  Measures: paper-pencil-assessment (last 7-d sedentary behavior questionnaire, SIT-Q-7d)
sedentary time by accelerometry | Change from Baseline Sedentary Time at 12 months
  Measures: objective measurement of physical activity by accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Ulbricht, Dr., Study Chair — Institute of Social Medicine and Prevention, University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Voigt L, Baumann S, Ullrich A, Weymar F, John U, Ulbricht S. The effect of mere measurement from a cardiovascular examination program on physical activity and sedentary time in an adult population. BMC Sports Sci Med Rehabil. 2018 Jan 23;10:1. doi: 10.1186/s13102-018-0090-8. eCollection 2018. PMID 29410786
- [Result] Ullrich A, Voigt L, Baumann S, Weymar F, John U, Dorr M, Ulbricht S. A cross-sectional analysis of the associations between leisure-time sedentary behaviors and clustered cardiometabolic risk. BMC Public Health. 2018 Mar 6;18(1):327. doi: 10.1186/s12889-018-5213-3. PMID 29510707
- [Result] Baumann S, Gross S, Voigt L, Ullrich A, Weymar F, Schwaneberg T, Dorr M, Meyer C, John U, Ulbricht S. Pitfalls in accelerometer-based measurement of physical activity: The presence of reactivity in an adult population. Scand J Med Sci Sports. 2018 Mar;28(3):1056-1063. doi: 10.1111/sms.12977. Epub 2017 Oct 12. PMID 28921747
- [Derived] Voigt L, Ullrich A, Gross S, Guertler D, Jaeschke L, Dorr M, van den Berg N, John U, Ulbricht S. Associations of accelerometer-based sedentary bouts with adiposity markers among German adults - results from a cross-sectional study. BMC Public Health. 2023 Mar 10;23(1):469. doi: 10.1186/s12889-023-15304-8. PMID 36899317
- [Derived] Voigt L, Ullrich A, Baumann S, Dorr M, John U, Ulbricht S. Do sociodemographic variables and cardiometabolic risk factors moderate the mere-measurement effect on physical activity and sedentary time? BMC Cardiovasc Disord. 2020 Jun 5;20(1):272. doi: 10.1186/s12872-020-01551-9. PMID 32503441